CLINICAL TRIAL: NCT06518655
Title: Exploratory Study on the Identification of Benign and Malignant Pulmonary Nodules Using Volatile Organic Compounds in Human Exhaled Breath
Brief Title: Differentiation of Benign and Malignant Pulmonary Nodules by Volatile Organic Compounds in Human Exhaled Breath
Status: Recruiting | Type: Observational
Sponsor: ChromX Health (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); First People's Hospital of Foshan (Other); Sichuan Cancer Hospital and Research Institute (Other); Liwan District Central Hospital (Unknown); Shanghai Chest Hospital (Other); Peking Union Medical College Hospital (Other); Guangzhou Development Zone Hospital (Unknown); Huangpu District Hongshan Street Community Health Service Center (Unknown); Huangpu District Chinese Medicine Hospital (Unknown); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Huangpu District Jiufo Street Community Health Service Center (Unknown); Huangpu District Xinlong Town Central Hospital (Unknown); Huangpu District Yonghe Street Community Health Service Center (Unknown); Huangpu District Lianhe Street Second Community Health Service Center (Unknown); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: LCLN01
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Nodules, Multiple; Pulmonary Nodules, Solitary; Lung Cancer
Keywords: Pulmonary Nodules; Lung Cancer; Volatile Organic Compounds; Human Exhaled Breath
MeSH Terms: conditions — Multiple Pulmonary Nodules; Solitary Pulmonary Nodule; Lung Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Volatile Organic Compounds in Human Exhaled Breath
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Nodules: Pre-surgery adult patients with pulmonary nodule found by CT scan.
  Interventions: Other: Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system

INTERVENTIONS:
Other: Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system — Detection of volatile organic compound molecules in human exhaled breath by GC-MS and μGC-PID

SUMMARY:
The goal of this observational study is to develop an advanced expiratory algorithm model utilizing exhaled breath volatile organic compound (VOC) markers. This model aims to accurately differentiate benign from malignant nodules in individuals harboring pulmonary nodules. The primary objectives it strives to accomplish are:

1. To assess the diagnostic accuracy of an exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model in distinguishing benign and malignant pulmonary nodules.
2. To evaluate the diagnostic effectiveness of an AI model that employs exhaled breath VOC biomakers to identify specific types of malignant nodules, including lung adenocarcinoma, lung squamous cell carcinoma, and small cell lung cancer.
3. To explore and identify key characteristic VOCs combinations that are associated with EGFR site mutations in malignant nodules, further modeling and evaluating the classification performance.

By utilizing this comprehensive approach, the study hopes to contribute significantly to early detection and accurate classification of pulmonary nodules, ultimately leading to improved patient care and treatment outcomes.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional, and observational cohort study aiming at recruiting 3000 participants with pulmonary nodules ranging from 5 to 30 mm in diameter. Prior to invasive surgery, exhaled breath samples will be collected from these participants and analyzed using Gas chromatography-mass spectrometry(GC-MS) and micro Gas Chromatography-photoionisation detector (μGC-PID) system. Following the acquisition of μGC-PID results, a comprehensive evaluation of the diagnostic performance of VOC biomakers distinguishing between benign and malignant pulmonary nodules will be conducted, leveraging histopathological findings, CT examination data, and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* Pulmonary nodules were detected through low-dose spiral CT, chest CT conventional scan, or high-resolution thin-layer CT examination, with a maximum diameter of 5-30 mm, including solid nodules and ground glass nodules;
* Patients require pulmonary nodule resection to define the type of nodule pathology;
* The Patients have not yet used any drugs for tumor treatment;
* Patients and/or family members are able to understand the research protocol and are willing to participate in this study, providing written informed consent.

Exclusion Criteria:

* The maximum diameter of pulmonary nodules is greater than 30 mm;
* Patients are unable to determine the pathological diagnosis of pulmonary nodules after surgical resection or biopsy;
* Patients with recurrent lung cancer;
* Patients who have undergone lung transplantation or lobectomy;
* Individuals who currently or have a history of malignant tumors;
* Patients in the acute phase of inflammation or in need of intensive care in the above selected disease groups;
* Individuals with severe liver and kidney dysfunction;
* Mental illness patients (such as severe dementia, schizophrenia, severe depression, manic depressive psychosis, etc.);
* Confirmed HIV patients;
* Pregnant or lactating women;
* Patients or family members are unable to understand the conditions and objectives of this study.
* The patient is unwilling or unable to personally sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have pulmonary nodules with a large diameter between 5 mm and 30 mm on a CT scan within six months.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of an exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model in distinguishing benign and malignant pulmonary nodules. | 3 years
  The diagnostic performance of the exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model will be compared with pathologic diagnosis and CT/LDCT data, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

SECONDARY OUTCOMES:
The diagnostic effectiveness of an AI model to identify specific types of malignant nodules, including lung adenocarcinoma, lung squamous cell carcinoma, and small cell lung cancer. | 3 years
  The diagnostic performance of the exhaled breath VOC-assisted diagnostic artificial intelligence (AI) model will be compared with pathologic diagnosis, including sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV).

OTHER OUTCOMES:
Establish an exhaled breath VOC model for predicting EGFR mutations in malignant pulmonary nodules. | 3 years
  Establish an exhaled breath VOC model for predicting EGFR mutations in pathologically confirmed malignant pulmonary nodules. And evaluate the prediction accuracy by comparing the results of EGFR gene testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (15):
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - First People's Hospital of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Liwan District Central Hospital, Guangzhou, Guangdong
  - Guangzhou Development Zone Hospital, Guangzhou, Guangdong
  - Huangpu District Chinese Medicine Hospital, Guangzhou, Guangdong
  - Huangpu District Hongshan Street Community Health Service Center, Guangzhou, Guangdong
  - Huangpu District Jiufo Street Community Health Service Center, Guangzhou, Guangdong
  - Huangpu District Lianhe Street Second Community Health Service Center, Guangzhou, Guangdong
  - Huangpu District Xinlong Town Central Hospital, Guangzhou, Guangdong
  - Huangpu District Yonghe Street Community Health Service Center, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Shlomi D, Abud M, Liran O, Bar J, Gai-Mor N, Ilouze M, Onn A, Ben-Nun A, Haick H, Peled N. Detection of Lung Cancer and EGFR Mutation by Electronic Nose System. J Thorac Oncol. 2017 Oct;12(10):1544-1551. doi: 10.1016/j.jtho.2017.06.073. Epub 2017 Jul 12. PMID 28709937
- [Background] van de Goor R, van Hooren M, Dingemans AM, Kremer B, Kross K. Training and Validating a Portable Electronic Nose for Lung Cancer Screening. J Thorac Oncol. 2018 May;13(5):676-681. doi: 10.1016/j.jtho.2018.01.024. Epub 2018 Feb 6. PMID 29425703
- [Background] Hanna GB, Boshier PR, Markar SR, Romano A. Accuracy and Methodologic Challenges of Volatile Organic Compound-Based Exhaled Breath Tests for Cancer Diagnosis: A Systematic Review and Meta-analysis. JAMA Oncol. 2019 Jan 1;5(1):e182815. doi: 10.1001/jamaoncol.2018.2815. Epub 2019 Jan 10. PMID 30128487
- [Background] Horvath I, Lazar Z, Gyulai N, Kollai M, Losonczy G. Exhaled biomarkers in lung cancer. Eur Respir J. 2009 Jul;34(1):261-75. doi: 10.1183/09031936.00142508. PMID 19567608
- [Background] Mitsui T, Kondo T. Inadequacy of theoretical basis of breath methylated alkane contour for assessing oxidative stress. Clin Chim Acta. 2003 Jul 1;333(1):91; author reply 93-4. doi: 10.1016/s0009-8981(03)00173-6. No abstract available. PMID 12809740
- [Background] Stone BG, Besse TJ, Duane WC, Evans CD, DeMaster EG. Effect of regulating cholesterol biosynthesis on breath isoprene excretion in men. Lipids. 1993 Aug;28(8):705-8. doi: 10.1007/BF02535990. PMID 8377584
- [Background] Nakhleh MK, Amal H, Jeries R, Broza YY, Aboud M, Gharra A, Ivgi H, Khatib S, Badarneh S, Har-Shai L, Glass-Marmor L, Lejbkowicz I, Miller A, Badarny S, Winer R, Finberg J, Cohen-Kaminsky S, Perros F, Montani D, Girerd B, Garcia G, Simonneau G, Nakhoul F, Baram S, Salim R, Hakim M, Gruber M, Ronen O, Marshak T, Doweck I, Nativ O, Bahouth Z, Shi DY, Zhang W, Hua QL, Pan YY, Tao L, Liu H, Karban A, Koifman E, Rainis T, Skapars R, Sivins A, Ancans G, Liepniece-Karele I, Kikuste I, Lasina I, Tolmanis I, Johnson D, Millstone SZ, Fulton J, Wells JW, Wilf LH, Humbert M, Leja M, Peled N, Haick H. Diagnosis and Classification of 17 Diseases from 1404 Subjects via Pattern Analysis of Exhaled Molecules. ACS Nano. 2017 Jan 24;11(1):112-125. doi: 10.1021/acsnano.6b04930. Epub 2016 Dec 21. PMID 28000444
- [Background] Zhou J, Huang ZA, Kumar U, Chen DDY. Review of recent developments in determining volatile organic compounds in exhaled breath as biomarkers for lung cancer diagnosis. Anal Chim Acta. 2017 Dec 15;996:1-9. doi: 10.1016/j.aca.2017.09.021. Epub 2017 Sep 13. PMID 29137702
- [Background] Arasaradnam RP, Wicaksono A, O'Brien H, Kocher HM, Covington JA, Crnogorac-Jurcevic T. Noninvasive Diagnosis of Pancreatic Cancer Through Detection of Volatile Organic Compounds in Urine. Gastroenterology. 2018 Feb;154(3):485-487.e1. doi: 10.1053/j.gastro.2017.09.054. Epub 2017 Nov 10. No abstract available. PMID 29129714
- [Background] Chan DK, Zakko L, Visrodia KH, Leggett CL, Lutzke LS, Clemens MA, Allen JD, Anderson MA, Wang KK. Breath Testing for Barrett's Esophagus Using Exhaled Volatile Organic Compound Profiling With an Electronic Nose Device. Gastroenterology. 2017 Jan;152(1):24-26. doi: 10.1053/j.gastro.2016.11.001. Epub 2016 Nov 5. No abstract available. PMID 27825962
- [Background] Gordon SM, Szidon JP, Krotoszynski BK, Gibbons RD, O'Neill HJ. Volatile organic compounds in exhaled air from patients with lung cancer. Clin Chem. 1985 Aug;31(8):1278-82. PMID 4017231
- [Background] Corradi M, Pesci A, Casana R, Alinovi R, Goldoni M, Vettori MV, Cuomo A. Nitrate in exhaled breath condensate of patients with different airway diseases. Nitric Oxide. 2003 Feb;8(1):26-30. doi: 10.1016/s1089-8603(02)00128-3. PMID 12586538
- [Background] Bousamra M 2nd, Schumer E, Li M, Knipp RJ, Nantz MH, van Berkel V, Fu XA. Quantitative analysis of exhaled carbonyl compounds distinguishes benign from malignant pulmonary disease. J Thorac Cardiovasc Surg. 2014 Sep;148(3):1074-80; discussion 1080-1. doi: 10.1016/j.jtcvs.2014.06.006. Epub 2014 Jun 8. PMID 25129599
- [Background] Phillips M, Altorki N, Austin JH, Cameron RB, Cataneo RN, Greenberg J, Kloss R, Maxfield RA, Munawar MI, Pass HI, Rashid A, Rom WN, Schmitt P. Prediction of lung cancer using volatile biomarkers in breath. Cancer Biomark. 2007;3(2):95-109. doi: 10.3233/cbm-2007-3204. PMID 17522431
- [Background] Phillips M, Bauer TL, Pass HI. A volatile biomarker in breath predicts lung cancer and pulmonary nodules. J Breath Res. 2019 Jun 19;13(3):036013. doi: 10.1088/1752-7163/ab21aa. PMID 31085817
- [Background] Phillips M, Cataneo RN, Greenberg J, Grodman R, Gunawardena R, Naidu A. Effect of oxygen on breath markers of oxidative stress. Eur Respir J. 2003 Jan;21(1):48-51. doi: 10.1183/09031936.02.00053402. PMID 12570108